CLINICAL TRIAL: NCT03912974
Title: Effects of Serotonin Transporter Inhibition on the Subjective Response to Psilocybin in Healthy Subjects
Brief Title: Effects of SERT Inhibition on the Subjective Response to Psilocybin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2019-00223
Record Dates: First submitted 2019-03-06; First posted 2019-04-12 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: 2-period cross-over, randomized, double-blinded (escitalopram vs. placebo)study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pretreatment condition is double-blinded (escitalopram 10 mg x 7 days, then 20 mg orally x 7 days vs. placebo (mannitol) orally x 14 days) On each of the 2 study days, participants will receive psilocybin 25 mg orally (no placebo control on the study days)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pretreatment with escitalopram (Active Comparator): Pretreatment with escitalopram (10 mg for 7 days orally, 20 mg for another 7 days orally), followed by administration of psilocybin (25 mg orally) on the study day
  Interventions: Drug: Escitalopram
- Pretreatment with placebo oral capsule (Placebo Comparator): Pretreatment with placebo, followed by administration of psilocybin (25 mg orally) on the study day
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Escitalopram — see 'arm description'
  Arms: Pretreatment with escitalopram
Drug: Placebo oral capsule — see 'arm description'
  Arms: Pretreatment with placebo oral capsule

SUMMARY:
Psilocybin is a classic serotonergic hallucinogen acting on the 5-HT2A receptor. It is used recreationally and in psychiatric research. Selective serotonin reuptake inhibitors (SSRIs) like escitalopram are first-line treatments for depression. They inhibit the serotonin transporter (SERT). This might cause a possible downregulation of postsynaptic 5-HT receptors, e.g. the 5-HT2A receptor. The aim of the study is to investigate the effects of psilocybin after escitalopram and Placebo pretreatment. Subjective and physiological effects as well as effects on gene expression will be assessed.

DETAILED DESCRIPTION:
Psilocybin (the active substance in "magic mushrooms") is a classic serotonergic hallucinogen acting on the serotonin 5-HT2A receptor. Psilocybin is used recreationally and in psychiatric research. First studies suggest efficacy in psychiatric disorders, such as depression. SSRIs like escitalopram are currently among the first-line treatments of this disorder. Escitalopram acts as a serotonin transporter (SERT) inhibitor. However, the link between this mechanism and its positive effects on mood remains to be established. Several studies suggest a possible downregulation of postsynaptic serotonin (5-HT) receptors such as the 5-HT2A receptor. The aim of the study is to assess whether SERT inhibition reduces expression of the gene coding for the 5-HT2A receptor and the response to psilocybin.

Participants will be treated with escitalopram (10 mg in the 1st and 20 mg in the 2nd week) or placebo for 14 days. Pretreatment is followed the first study day. A single dose of psilocybin (25 mg) will be administered. Primary study endpoint are the subjective effects on consciousness (measured by the 5D-ASC total score). Secondary study endpoints include additional psychological measurements, plasma concentrations of psilocybin and escitalopram, hydroxytryptamine receptor (HTR) gene expression, as well as some safety measures (autonomic effects, ECG). The washout between the first study day and the second pretreatment will be at least 2 days. In the second pretreatment period, participants will be treated with placebo or escitalopram (cross-over) for another 14 days. This is followed by the second study day and administration of psilocybin (25 mg).

Based on a power analysis the sample size is 24 participants (12 female and 12 male).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years.
2. Understanding of the German language.
3. Understanding the procedures and the risks that are associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 24 h after substance administration.
8. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session.
9. Women of childbearing potential must be willing to use double-barrier birth control.

Exclusion Criteria:

1. Chronic or acute medical condition, including a history of seizures.
2. Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders, and substance abuse).
3. Psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
4. Illicit substance use (with the exception of cannabis) more than 10 times or any time within the previous two months.
5. History of an angle closure glaucoma.
6. Pregnant or nursing women.
7. Participation in another clinical trial (currently or within the last 30 days).
8. Use of medications that may interfere with the effects of the study medications (any psychiatric medications and any medication with known pharmacokinetic or pharmacodynamic interactions with escitalopram).
9. A corrected QT time (QTc), calculated by Bazett's formula, of over 450 milliseconds in males and over 470 milliseconds in females.
10. Tobacco smoking (>10 cigarettes/day).
11. Consumption of alcoholic drinks (>10 drinks / week).
12. Bodyweight < 45 kg.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
5 dimensions of altered state of consciousness (5D-ASC) profile total score | 20 Months
  Visual analog scale consisting of 94 items. Constructed of five scales and allows assessing mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. Scales will be presented as 100 mm long horizontal lines marked with vertical lines by the participant.

SECONDARY OUTCOMES:
Visual Analog Scales (VAS) | 20 Months
  VAS will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS will be used: "any effect", "good effect", "bad effect","liking", "high", "happy", "fear", "stimulated", "feeling close to others", "concentration", "thinking", "open", "trust", "want to be with other people", "loss of sense of time", and "the boundaries between myself and my surroundings seemed to blur". Subjects will mark the scale with vertical lines.
Adjective mood rating scale (AMRS) | 20 Months
  The adjective mood rating scale (AMRS or EWL60S) is a 60-item Likert scale that allows repeated assessment of mood in 6 dimensions: activation, inactivation, well-being, anxiety/depressed mood, extroversion and introversion, and emotional excitability.The AMRS consists of subscales measuring "activation", "positive mood", "extroversion", "introversion", "inactivation", and "emotional excitability.
States of consciousness questionnaire (SCQ) | 20 Months
  This 100-item questionnaire is rated on a six-point scale. Forty-three items embedded into this questionnaire comprise the Mystical Experience Questionnaire (MEQ). which is sensitive to the effects of psilocybin. The 43 items provide scale scores for each of seven domains of mystical experiences: internal unity (pure awareness, a merging with ultimate reality), external unity (unity of all things, all things are alive, all is one), sense of sacredness (reverence, sacred), noetic quality (encounter with ultimate reality, more real than everyday reality), transcendence of time and space, deeply felt positive mood (joy, peace, love), paradoxicality/ineffability (claim of difficulty in describing the experience in words). We will also derived the four scale scores of the newly validated revised 30-item MEQ: mystical, positive mood, transcendence of time and space, and ineffability.
Mysticism scale (MS) | 20 Months
  The MS is a 32-item questionnaire that was developed to assess primary mystical experiences. The items are rated on a 9-point Likert scale. The scale consists of 16 positively worded statements and 16 negatively worded statements.
Eppendorf Schizophrenia Inventory (ESI) | 20 Months
  The ESI yields four schizophrenia-specific dimensions: attention and speech impairment (AS), ideas of reference (IR), auditory uncertainty (AU), and deviant perception (DP).
Blood pressure | 20 Months
  Repeatedly measured using blood pressure / pulse apparatus (mmHg scale)
Heart rate | 20 Months
  Repeatedly measured using blood pressure / pulse apparatus (beats per minute scale)
Body temperature | 20 Months
  Repeatedly measured using ear thermometer (degree Celsius scale)
Pupil diameter | 20 Months
  Repeatedly measured using pupil distance meter (millimeter scale)
Plasma concentrations of escitalopram | 20 Months
  Escitalopram plasma concentrations will be measured repeatedly over time using LC-MS/MS techniques (nanogram per milliliter scale)
Plasma concentrations of psilocin | 20 Months
  Escitalopram plasma concentrations will be measured repeatedly over time using LC-MS/MS techniques (nanogram per milliliter scale)
HTR gene expression | 20 Months
  Messenger ribonucleic acid (mRNA) expression levels in whole blood as a peripheral marker of spiny neuronal gene (CNS) expression will be used to measure expression of HTR genes as well as expression of the SERT gene.
Changes in the electrocardiogram (ECG) | 20 Months
  12-lead electrocardiogram will be measured twice on the study days (baseline and at peak drug effect) as well as on the screening exam to examine possible drug-induced changes in the ECG as well as a safety measure (millisecond scale).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Holze F, Becker AM, Kolaczynska KE, Duthaler U, Liechti ME. Pharmacokinetics and Pharmacodynamics of Oral Psilocybin Administration in Healthy Participants. Clin Pharmacol Ther. 2023 Apr;113(4):822-831. doi: 10.1002/cpt.2821. Epub 2022 Dec 31. PMID 36507738
- [Derived] Becker AM, Holze F, Grandinetti T, Klaiber A, Toedtli VE, Kolaczynska KE, Duthaler U, Varghese N, Eckert A, Grunblatt E, Liechti ME. Acute Effects of Psilocybin After Escitalopram or Placebo Pretreatment in a Randomized, Double-Blind, Placebo-Controlled, Crossover Study in Healthy Subjects. Clin Pharmacol Ther. 2022 Apr;111(4):886-895. doi: 10.1002/cpt.2487. Epub 2021 Nov 22. PMID 34743319